CLINICAL TRIAL: NCT06946901
Title: The Safety and Effectiveness of Hyperthermic Intraperitoneal Chemotherapy Combined With Intravenous Chemotherapy for Peritoneal Metastatic Pancreatic Cancer, a Phase II Clinical Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSPAC-09
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Hyperthermic Intraperitoneal Chemotherapy; Peritoneal Metastatic Pancreatic Cancer
MeSH Terms: interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HIPEC + AG Chemotherapy Group (Experimental)
  Interventions: Combination Product: Hyperthermic Intraperitoneal Chemotherapy (HIPEC) with Cisplatin + Systemic AG Chemotherapy

INTERVENTIONS:
Combination Product: Hyperthermic Intraperitoneal Chemotherapy (HIPEC) with Cisplatin + Systemic AG Chemotherapy — * HIPEC (cisplatin 70mg/m², Day 1,3 post-surgery), 1 cycle；
  * Systemic AG chemotherapy (nab-paclitaxel 125mg/m²+ gemcitabine 1000mg/m², initiated, Day 1,8,15, q4 week), 4 cycles

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness and safety of hyperthermic intraperitoneal chemotherapy combined with intravenous chemotherapy in peritoneal metastatic pancreatic cancer. The main question it aims to answer are:

(1) Does this combined approach increase 1-year survival rates? and (2) What is the safety profile of this treatment regimen?

Participants will:

undergo baseline imaging and surgical exploration to confirm peritoneal metastasis, receive two cycles of intraperitoneal cisplatin HIPEC (70mg/m²) postoperatively, followed by systemic AG chemotherapy (nab-paclitaxel plus gemcitabine), with treatment adjustments based on regular imaging assessments and multidisciplinary team (MDT) recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Obtain signed informed consent from the patient or their legal representative, with adherence to the study protocol and follow-up procedures;
* Aged >=18 and <=80 years, regardless of gender;
* No contraindications to surgery, with an ECOG performance status of 0-1;
* Confirmed peritoneal metastasis by imaging or intraoperative detection, with rapid intraoperative histopathology indicating metastatic adenocarcinoma;
* No prior anti-tumor therapy before treatment, including systemic chemotherapy, interventional chemotherapy, high-intensity focused ultrasound (HIFU), radiotherapy, immunotherapy, molecular targeted therapy, or traditional Chinese medicine anti-tumor treatments;
* No severe hematological, cardiac, pulmonary dysfunction, or autoimmune deficiency (based on respective diagnostic criteria);
* Hematological criteria: White blood cells (WBC) >=3.0 × 10⁹/L; Absolute neutrophil count (ANC) >=1.5 × 10⁹/L; Platelets (PLT) >=100 × 10⁹/L; Hemoglobin (Hgb) >=90 g/L.
* Blood biochemistry criteria: AST (SGOT) and ALT (SGPT) <=2.5 × upper limit of normal (ULN); Total bilirubin (TBIL) <=2 × ULN; Serum creatinine (CRE) <=1.5 × ULN.
* Coagulation function: Prothrombin time (PT) and international normalized ratio (INR) <=1.5 × ULN;
* Compliance with study visit schedules and other protocol requirements.

Exclusion Criteria:

* Presence of distant metastases to other organs (e.g., liver, bone, lung) with definitive evidence, except for ovarian metastases;
* History of other systemic malignancies within the past five years;
* Use of any non-anti-tumor investigational drugs within 4 weeks prior to treatment;
* Accompanied by massive ascites (extending from pelvic to upper abdominal cavity);
* History of upper gastrointestinal bleeding requiring repeated blood transfusions within the past three months;
* Pregnancy, autoimmune diseases, severe hyperthyroidism/hypothyroidism, central nervous system disorders, psychiatric illnesses, unstable angina, congestive heart failure, severe arrhythmias, or other uncontrolled serious medical conditions;
* History of hypersensitivity to the study drugs or medications with similar chemical structures;
* Patients requiring long-term warfarin anticoagulation therapy;
* Poor compliance, inability or unwillingness to provide signed informed consent;
* Patients likely to be lost to follow-up for ≥14 days during the treatment period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-04-03 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year Overall Survival (OS) Rate | From enrollment to 12 months post-treatment initiation
  The proportion of patients alive at 12 months after initiation of the combined HIPEC and systemic AG chemotherapy treatment, analyzed by Kaplan-Meier method.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From enrollment until first documented progression or death (up to 24 months)
  Time from treatment initiation to radiographic disease progression (per RECIST 1.1) or death from any cause, whichever occurs first, assessed by blinded independent central review (BICR).
Objective Response Rate (ORR) | From enrollment until end of treatment (up to 12 months)
  Proportion of patients achieving complete response (CR) or partial response (PR) per RECIST 1.1 criteria during the study intervention period.
Safety and Tolerability (CTCAE v5.0) | From first HIPEC cycle to 30 days after last treatment (up to 13 months)
  Frequency and severity of adverse events (AEs), serious AEs (SAEs), and treatment discontinuations due to AEs, graded by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality